CLINICAL TRIAL: NCT00115154
Title: Vehicle-Controlled, Double-Blind Study to Assess the Safety and Efficacy of Imiquimod 5% Cream for the Treatment of Actinic Keratosis on the Upper Extremities
Brief Title: Study to Assess the Safety and Efficacy of Imiquimod 5% Cream for the Treatment of Actinic Keratosis on the Arms and Hands
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Graceway Pharmaceuticals, LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1516-IMIQ
Record Dates: First submitted 2005-06-21; First posted 2005-06-22 (Estimated); Last update posted 2007-02-19 (Estimated); Status verified 2007-02

CONDITIONS: Keratosis
Keywords: Actinic Keratosis; AK; 3M Pharmaceuticals; Aldara; Imiquimod; Actinic Keratosis (AK)
MeSH Terms: conditions — Keratosis; Keratosis, Actinic | interventions — Imiquimod

INTERVENTIONS:
Drug: Aldara (imiquimod) cream, 5%

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of imiquimod 5% cream compared to vehicle cream in the treatment of Actinic Keratosis (AK) on the arm and/or hand when the cream is applied once daily 2 days per week for 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Have AK on arm or hand
* Discontinuation of sun tanning and the use of tanning beds
* Discontinuation of the use of moisturizers, body oils, over-the-counter retinol products and products containing alpha or beta hydroxy acid in the treatment and surrounding area
* Withholding of the use of sunscreen in the treatment area for 24 hours prior to all study visits and for 8 hours before applying study cream
* Postponement of the treatment of non-study AK lesions anywhere on the arm being treated until study participation is complete

Exclusion Criteria:

* Subjects must not have any evidence of systemic cancer or immunosuppression or other unstable health conditions
* Participation in another clinical study
* Have previously received treatment with imiquimod within the treatment area
* Have squamous cell carcinoma (SCC), basal cell carcinoma (BCC), or other malignancy in the treatment or surrounding area that requires treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 270
Dates: Start 2005-05; Study Completion 2006-09

PRIMARY OUTCOMES:
The primary objective of this study is to evaluate the efficacy of imiquimod 5% cream compared to vehicle cream in the treatment of AK on the upper extremities when the cream is applied once daily 2 days per week for 16 weeks.

SECONDARY OUTCOMES:
The secondary objective is to evaluate the safety of treatment with imiquimod 5% cream in subjects with AK lesions on the upper extremities.

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Tucson, Arizona
  - Vista, California
  - Atlanta, Georgia
  - Newnan, Georgia
  - Buffalo Grove, Illinois
  - Evansville, Indiana
  - Riverside Park, New Jersey
  - New York, New York
  - Rochester, New York
  - Greenville, North Carolina
  - Portland, Oregon
  - Providence, Rhode Island
  - Knoxville, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - Virginia Beach, Virginia
  - Wenatchee, Washington
  - Milwaukee, Wisconsin